CLINICAL TRIAL: NCT02074670
Title: FUNCTIONAL MAGNETIC RESONANCE IMAGING (fMRI) OF THE SENSORIMOTOR CORTEX IN SPINAL CORD INJURY PATIENT AFTER INTENSIVE REHABILITATION INCLUDING ROBOTIC DEVICES
Brief Title: fMRI In Spinal Cord Injury Patient After Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade do Vale do Paraíba (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Professor, University of Nove de Julho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL003
Record Dates: First submitted 2014-02-17; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treadmill gait training (Experimental): Five days a week, 40 sessions of Kinesiotherapy (passive and active mobilizations, muscle lengthening), Body Weight Supported Treadmill Training, bicycle, manual therapy (with and without assistance of a mechanical device) and daily life activities training.
  Interventions: Other: Treadmill gait training

INTERVENTIONS:
Other: Treadmill gait training — Five days a week, 40 sessions of Kinesiotherapy (passive and active mobilizations, muscle lengthening), Body Weight Supported Treadmill Training, bicycle, manual therapy (with and without assistance of a mechanical device) and daily life activities training.

SUMMARY:
The purpose of this study was to evaluate the potential reorganization in the sensorimotor cortex in spinal cord injury (SCI) patients after Body Weight Supported Treadmill Training (BWSTT) associated with conventional motor rehabilitation. The investigators hypothesized that training with weight bearing associated with conventional motor rehabilitation will be able to reorganize the brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASIA C or D and the ability to cooperate with instructions of the motor task required. The motor task was to perform ankle plantar flexion and toe flexion and fingers and thumbs movement of the both sides; they also had to be able to fulfill the general conditions necessary for an MRI exploration.

Exclusion Criteria:

* Patients with uncontrollable spasticity-induced body movements were excluded from the study.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Cortical Motor Area | 1 month
  Cortical Motor area in fMRI during motor task.

SECONDARY OUTCOMES:
Functional Index | 1 month
  Walking Index for Spinal Cord Injury

CONTACTS AND LOCATIONS:
Locations (1):
- Paulo Roberto Garcia Lucareli, São Paulo, São Paulo, Brazil